CLINICAL TRIAL: NCT03146832
Title: Exposure Works, But How? Testing Different Therapeutic Strategies During Exposure to Pain in an Experimental Design
Brief Title: Therapeutic Strategies During Exposure to Pain in an Experimental Design
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Philipps University Marburg (Other)
Responsible Party: Principal Investigator, Julia Anna Glombiewski, Ph.D, Licensed Psychologist, Principal Investigator, Philipps University Marburg
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2016-33v
Record Dates: First submitted 2017-04-18; First posted 2017-05-10 (Actual); Last update posted 2017-07-05 (Actual); Status verified 2017-07

CONDITIONS: Pain, Acute
MeSH Terms: conditions — Acute Pain | interventions — Implosive Therapy

STUDY DESIGN:
Intervention Model Description: participants are assigned to one of three experimental groups in parallel for the duration of the study
Who Masked: Participant
Masking Description: Participants were not aware which experimental condition they were allocated to.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Habituation (Experimental): The habituation instruction focuses on changes of the initial physical fear-responses during exposure sessions. It is explained that the level of anxiety will gradually decrease, or habituate, each time someone faces a feared situation. Participants are then instructed to observe their own level of fear during the three practice trials with the thermode. Together with the experimenter, participants have to indicate their level of arousal on an 11-point scale (0= neutral, 10 = very high) in-between and after the three practice trials. After the practice trial, participants are instructed to reconsider their own development of physical responses. Participants are encouraged to remember the development of their level of arousal during the test trail with the thermode.
  Interventions: Behavioral: Exposure therapy (according to habituation approach)
- Expectation Violation (Experimental): The expectation violation instruction focuses on the verification of negative expectancies during exposures sessions. It is explained that exposure exercises help to create own experiences which allow to directly test negative predicted outcomes. Together with the experimenter, participants are then encouraged to formulate concrete concerns in regard to the practice trail with the thermode. Before the practice trails, participants have to indicate the likelihood of their concerns on an 11-point scale (0= not likely, 10 = very likely). After the practice trails, participants are instructed to evaluate their own concerns by some guided questions (e.g. "What did you learn?"). Participants are encouraged to keep their own experience in mind during the test trail with the thermode.
  Interventions: Behavioral: Exposure therapy (according to inhibitory learning approach)
- Control (No Intervention): Participants in the control group are not provided with information about exposure therapy. Instead, participants listen to a newspaper article which reports on the daily work in a botanical garden. Together with the experimenter, participants are then asked to name the most interesting aspect in the article. Before the practice trails, participants have to rate how likely it is that they would further inform themselves about botanical gardens on an 11-point scale (0= not likely, 10 = very likely). After the practice trails, participants are provided with some further questions about the newspaper article (e.g. "Did you find the newspaper article interesting?"). This cognitive exercise does not cover any pain-related topics and, therefore, does not serve as a distraction instruction.

INTERVENTIONS:
Behavioral: Exposure therapy (according to habituation approach) — Exposure instruction focuses on fear reduction during exposure sessions
  Arms: Habituation
Behavioral: Exposure therapy (according to inhibitory learning approach) — Exposure instruction focuses on expectation violation during exposure sessions
  Arms: Expectation Violation

SUMMARY:
The goal of the present study is to compare different therapeutic strategies (according to habituation model vs. according to the inhibitory learning approach) during exposure to thermal pain in an experimental design.

DETAILED DESCRIPTION:
Exposure therapy is effective for the treatment of individuals with chronic pain and high levels of fear-avoidance. Nevertheless, mechanisms of change for exposure treatment are not sufficiently investigated. According to the habituation model, the activation of a fear structure leads to a habituation of the initial physical response. Therefore, the therapeutic recommendation is to focus on the reduction of fear during exposure sessions. According to the inhibitory learning approach, however, exposure experiences compete with the original US-CS fear association. Therefore, the therapist should maximize the violation of negative expectancies. The present study intends to compare both strategies during the exposure to pain in an experimental design.

ELIGIBILITY:
Inclusion Criteria:

* female gender
* sufficient knowledge of German language

Exclusion Criteria:

* chronic and acute pain conditions
* Raynaud's disease
* high blood pressure
* neuropathy, coronary diseases
* diabetes, current alcohol
* drug or pain-medication (last 24hours)

Ages: 18 Years to 60 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 139 (Actual)
Dates: Start 2017-04-01 (Actual); Primary Completion 2017-06-15 (Actual); Study Completion 2017-06-15 (Actual)

PRIMARY OUTCOMES:
Pain tolerance | 5 minutes prior and 5 minutes after three exposure practice trials
  Determined by the temperature at which the participant stopped the heat stimulus

SECONDARY OUTCOMES:
Pain intensity | 5 minutes prior and 5 minutes after three exposure practice trials
  Measured on an 11-point scale (0 = no pain; 10 = worst imaginable pain)
Pain quality | 5 minutes prior and 5 minutes after three exposure practice trials
  Measured on an 11-points scale (0 = bearable; 10 = unbearable)
Pain Catastrophizing Scale (PCS) | 1-week prior and 10 minutes after three exposure practice trials
  Pain catastrophizing thoughts (e.g. "I worry all the time about whether the pain will end.")
Pain Anxiety Symptom Scale (PASS) | 1-week prior and 10 minutes after three exposure practice trials
  Pain-related anxiety (e.g. "I worry when I am in pain.")
Pain Processing (Fragebogen zur Erfassung der Schmerzverarbeitung, FESV) | 1-week prior and 10 minutes after three exposure practice trials
  Cognitive pain coping strategies (e.g. "When I am in pain, I know several possibilities how to handle them.")
Psychophysiological activation | throughout the experiment (5 minutes prior, during and 10 minutes after three exposure practice trails
  e.g. skin conductance responses, heart rate

CONTACTS AND LOCATIONS:
Overall Officials: Julia Anna Glombiewski, Phd, Principal Investigator — Department of Clinical Psychology and Psychotherapy
Locations (1):
- Philipps University Marburg, Department of Clinical Psychology and Psychotherapy, Marburg, Germany

IPD SHARING:
Plan to Share IPD: No